CLINICAL TRIAL: NCT02235012
Title: Cognitive Biases in Decision Making in a Pharmacological Model of Psychosis : a Study in Healthy Humans Recieving Low Dose Anesthetic, Ketamine Versus Placebo
Brief Title: Cognitive Biases Under Ketamine
Acronym: KETABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Fondation pour la Recherche Médicale (Other); Fondation Fyssen (Unknown); Comité pour la Recherche Hospitalière Médicale (Unknown); Association Schizo Oui (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D512; 2013-002056-33 (EudraCT Number)
Record Dates: First submitted 2014-08-12; First posted 2014-09-09 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Healthy Subjects
Keywords: Schizophrenia; Ketamine; Cognitive biases; Uncertainty
MeSH Terms: conditions — Schizophrenia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine then placebo (Experimental): Infusion of low dose Ketamine then infusion of a saline solution
  Interventions: Drug: Ketamine; Drug: Placebo
- Placebo then ketamin (Experimental): Infusion of a saline solution then infusion of low dose Ketamine
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — KETAMINE PANPHARMA 250 mg/5mL, solution for infusion :
  * Initial rapid infusion of 0,23 mg/kg
  * Infusion from minute 2 to minute 30 : 0,00967 mg/kg/min
  * Infusion from minute 31 to minute 120 : 0,00483 mg/kg/min
Drug: Placebo — CHLORURE DE SODIUM 0,9 % MACOPHARMA :
  * Initial rapid infusion of 0,23 mg/kg
  * Infusion from minute 2 to minute 30 : 0,00967 mg/kg/min
  * Infusion from minute 31 to minute 120 : 0,00483 mg/kg/min

SUMMARY:
Characterise cognitive biases resulting from low dose ketamine infusion, used as a pharmacological model of psychosis.

Our assumption is that low dose ketamine results in reasoning biases by impairing the way uncertainty is monitored and taken into account for decision making.

DETAILED DESCRIPTION:
Ketamine is a non-competitive glutamate NMDA antagonist. The infusion of subanesthetic doses of ketamine results in sub-clinical schizophrenia-like positive symptoms in healthy controls. The safety of ketamine use is attested by its daily use in child anesthesia and by a number of studies showing there is no medical, neural or cognitive complication after a single infusion.

Low dose ketamine is therefore a valid and safe human model to study psychosis. The objective of the study is to characterise cognitive biases resulting from low dose ketamine infusion, used as a pharmacological model of psychosis.

We designed four distinct paradigms designed to better characterize these biases.

P1 is a neuroeconomic task where subjects have to make binary choices to maximize gains, in a situation where either direct feedback information or additional counterfactual information is provided.

P2 is a neuroeconomic task where a direct manipulation of uncertainty is performed, and its impact on decision is measured.

P3 is a perceptual decision making task, where subjects have to classify a gabor orientation into the diagonal or cardinal category based on a rapidly presented series of individual gabors. The contribution of each piece of evidence to the final decision is measured and correlated to fluctuations in eeg data.

P4 is a perceptual decision making task, where subjects have to determine the global orientation of a series of sequentially presented gabor stimulus. There are interim responses and final responses, the influence of the former on the latter (confirmation bias) is studied.

Our assumption is that low dose ketamine results in reasoning biases by impairing the way uncertainty is monitored and taken into account for decision making.

The study design is as follows : randomized, double blind, controlled, against placebo, cross-over.

Healthy subjects will therefore be randomized to receive on the first visit either a ketamine infusion or a placebo infusion. The alternative condition will be applied on the second visit.

Ketamine will be prepared using KETAMINE PANPHARMA 250 mg/5mL, and infusion will be. This procedure should produce ketamine plasmatic levels of 140ng/ml. Two blood samples will be taken 30 and 90 minutes after infusion start to record actual ketamine plasmatic levels.

Placebo infusion will follow the same pattern of infusion, prepared using CHLORURE DE SODIUM 0,9% MACOPHARMA.

We will record both behavioral, electrophysiologic and psychometric data. Detailed assumptions are as folllows :

Behavioral data :

P1 and 2 : Significant impairment with ketamine in the ability to take into account uncertainty to guide decisions.

P3 : Significant decrease with ketamine in the ability to classify correctly the mean spatial orientation of stimuli according to the cardinal or diagonal direction.

P4 : Significant increase with ketamine in the confirmation bias following the interim choice.

Electroencephalographic data :

Correlation between the impairment in the ability to take into account uncertainty and the alteration of the Error Related Negativity and late inhibitory eeg signals, and decreased long distance synchrony as indicated by spectral analysis (P1 and 2).

The covariation of brain activity with the weight each stimuli sample will have in the final decision, will be increased as a result of ketamine infusion (P3).

Psychometric data :

Increase in the Brief Psychiatric Rating Scale (BPRS) as a result of ketamine infusion. The BPRS scale records the psychotic symtoms and is translated and validated in a french population sample.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (as assessed by the Edinburgh scale)
* Aged 18 to 39
* Having given an informed consent
* Health insurance

Exclusion Criteria:

* Pregnant or breastfeeding woman (a urine pregnancy test will be offered in doubt)
* Personal or first-degree family history of psychosis
* Personal history of mood disorder, anxiety disorder, obsessive-compulsive disorder, somatoform disorder, dependence on a psychoactive substance, behavior disorder incompatible with a 2 hours EEG recording.
* Psychotropic treatment, current or stopped for less than 1 month, including antidepressant, anxiolytic but excluding hypnotic treatments.
* Personal history of neurologic disorder in relation to the central nervous system : congenital malformation of the brain, brain tumor, multiple sclerosis, degenerative disease of the central nervous system, epilepsy, current or in remission for less than 3 years or still requiring a medical treatment, inflammatory disease of the central nervous system dating under a year or having resulted in sequelae.
* Known hypertension or blood pressure above 140/90 mmHg upon clinical examination, congenital heart disease, ischemic heart disease, cardiac insufficiency, supraventricular and ventricular heart rhythm disorder.
* Person with restricted liberty, as a result of judicial or administrative measures
* Persons under involuntary commitment as a result of a psychiatric disorder.
* Person subject to a measure of legal protection or unable to consent.
* Known intolerance ketamine.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Evidence for biaises in decision making in an uncertain environment. | During infusion of Ketamine / Placebo (expected 2 hours)
  Behavioural analyses of decision making during the neuroeconomic or perceptual decision makin tasks (Paradigms 1 to 4)

SECONDARY OUTCOMES:
Electroencephalographic data | During infusion of Ketamine / Placebo (expected 2 hours)
  Correlation between the impairment in the ability to take into account uncertainty and the alteration of the Error Related Negativity and late inhibitory eeg signals, and decreased long distance synchrony as indicated by spectral analysis (Paradigms 1 and 2).
  The covariation of brain activity with the weight each stimuli sample will have in the final decision, will be increased as a result of ketamine infusion (Paradigm 3)
Brief Psychiatric Rating Scale (BPRS) | 30 and 90 minutes after infusion onset
Heart rate | Every 15 minutes during infusion
Pulse oxymetry | Every 15 minutes during infusion
Blood pressure | Every 15 minutes during infusion
Clinician administred dissociatives states scales (CADSS) | 30 and 90 minutes after infusion onset

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël GAILLARD, Principal Investigator — Centre Hospitalier St Anne
Locations (1):
- Centre Hospitalier Sainte Anne, Paris, France